CLINICAL TRIAL: NCT00528827
Title: A Randomized, Double-blinded, Placebo-controlled, Dose-ranging Study of Cardene® I.V. in Pediatric Subjects With Hypertension
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the sale of Cardene IV, the sponsor has stopped enrollment and withdrawn the study. No safety issues were identified.
Sponsor: Facet Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cardene® I.V. 1406
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Hypertension
Keywords: Hypertension, High Blood Pressure, Pediatric Hypertension, High blood pressure in children
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Drug: Cardene® I.V.
- 2 (Experimental): 5 mcg
  Interventions: Drug: Cardene® I.V.
- 3 (Experimental): 2.5
  Interventions: Drug: Cardene® I.V.
- 4 (Experimental): 0.5
  Interventions: Drug: Cardene® I.V.

INTERVENTIONS:
Drug: Cardene® I.V. — * 5 mcg/kg/min Cardene I.V.
  * 2.5 mcg/kg/min Cardene I.V.
  * 0.5 mcg/kg/min Cardene I.V.

SUMMARY:
To define the relationship between Cardene I.V. dose, serum concentrations, and blood pressure reduction in pediatric subjects with hypertension.

DETAILED DESCRIPTION:
Children with acute hypertensive episodes are frequently treated with the same marketed drugs as adults. Few drugs are specifically indicated for use in children with severe hypertension. Cardene I.V. has been widely used in children with severe hypertension without specific dosing recommendations for children in the labeling. This study is designed to examine the pharmacokinetics, pharmacodynamics, safety, and efficacy of using Cardene I.V. to reduce blood pressure (BP) in children with hypertension and will provide important information to guide use in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of Stage 1 or Stage 2 systolic hypertension at the time of screening.
* Male or female subjects, ages ≥2 to ≤16 years.
* Females who meet either of the following criteria:

  * Non-childbearing potential , as documented by:

    1. a medical history of non-menstruation or
    2. surgical sterility from oophorectomy and/or hysterectomy. * A history of tubal ligation or evidence of a sterile sexual partner is insufficient evidence of non-childbearing potential.
  * Childbearing potential: provide a negative urine pregnancy test within 24 hours of administration of study drug and agree to utilize effective contraception or remain abstinent during the entire treatment and follow-up periods of the study.
* Signed informed consent provided by an authorized subject representative and assent from subject, if feasible (based on local Institutional Review Board (IRB)/ethics panel requirements).

Exclusion Criteria:

* Subjects with seizures, altered state of consciousness, chest pain, facial palsy or intracranial hemorrhage at the time of screening.
* Receiving antihypertensive medication within a duration specified prior to screening.
* Treatment with cimetidine within 10 hours prior to dosing with study drug.
* Any known or suspected allergy to nicardipine hydrochloride.
* A calculated Glomerular Filtration Rate (GFR) under 30 mL/min/ 1.73 m2 as calculated using the Schwartz formula and the associated K values.
* Known history of severe aortic stenosis.
* Known history of severe left ventricular dysfunction.
* Known history of severely impaired hepatic function with portal hypertension.
* Liver function test (AST or ALT) results greater than or equal to twice the upper limit of normal.
* Receiving maintenance hemodialysis at screening or anticipated to require hemodialysis within 12 hours following initiation of treatment with study drug.
* Receiving a blood transfusion at screening or anticipated to require blood transfusions within 12 hours following initiation of treatment with study drug.
* Lack of appropriate intravenous (I.V.) access.
* Inability to tolerate a large-volume I.V. infusion.
* Any other condition or prior therapy, which, in the opinion of the investigator, would make the subject unsuitable for this study.
* Participation in any phase of another clinical research study involving the evaluation of another investigational drug or device within 30 days before randomization.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Mean percent change in SBP (Systolic Blood Pressure) from baseline during the 30-minute Randomized, Placebo-controlled Infusion Phase for each dose level of Cardene I.V. compared to placebo. | 30 minutes

SECONDARY OUTCOMES:
1) Mean percent change in SBP and DBP between various phases of dosing. 2) Proportion of subjects requiring additional antihypertensive medications during the treatment period. 3) Mean effective dose of Cardene I.V. | 72

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Beverly Hills, California
  - Miami, Florida